CLINICAL TRIAL: NCT00588328
Title: The Use of Breathing Synchronized CT and PET Scans in Radiation Therapy Treatment Planning
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00-008
Record Dates: First submitted 2007-12-20; First posted 2008-01-08 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Lung Cancer; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lung Neoplasms; Lymphoma, Non-Hodgkin | interventions — Positron Emission Tomography Computed Tomography

ARMS (1):
- 1 (Experimental)
  Interventions: Device: PET/CT scan

INTERVENTIONS:
Device: PET/CT scan — PET/CT scans

SUMMARY:
The purpose of this study is to find out whether a new device can help obtain more accurate CT and PET scans of the lungs and chest tumors and the liver and liver tumors to help in delivering radiation therapy. When we breathe, the amount of air in the lung changes. Lung tumors may also move during breathing. Liver tumors may also move with breathing; as the lungs inflate, the liver can be pushed down. A CT scan (a special type of X-ray) is routinely obtained as part of planning for lung or liver radiation therapy. Since patients breathe during this CT scan and their lung or liver tumors move, these CT scans can sometimes be inaccurate. We are now testing a device to only obtain the CT and an additional PET scan while patients are breathing in or out. This will hopefully allow us to deliver radiation with more accuracy.

DETAILED DESCRIPTION:
The objectives are to measure the amount of tumor motion with respiration, measure changes in tumor definition with breathing synchronized PET compared to standard free breathing PET, and to determine the fraction of patients whose radiation treatment plans would be modified based on this information. Eligible patients are those receiving radiation treatment for thoracic or liver tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Ability to sign informed consent form indicating investigative nature of this study, in keeping with the policies of the hospital.
* Patients must have thoracic disease visible on a Chest CT scan, or liver disease visible on a abdominal CT scan.

Exclusion Criteria:

* Pregnant women are ineligible. A pregnancy test will be performed on each fertile premenopausal female prior to entry into the study.
* Patients with thoracic or liver disease that is not visible on CT scan
* Patients who are unable to follow directions either due to language difficulties or hearing impairment.
* Patients who are too ill to hold their breath.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2000-03; Primary Completion 2008-07 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To measure the amount of tumor motion in breathing synchronized CT scans and determine the fraction of patients whose radiation treatment planning margins would be modified based on this information. | 2 years

SECONDARY OUTCOMES:
To measure changes in tumor definition with breathing synchronized PET compared to standard free breathing PET, and determine the fraction of patients whose radiation treatment plans would be modified based on this information. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Rosenzweig, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org